CLINICAL TRIAL: NCT04778722
Title: Development of Microbiome Vaginae After Use of Oral Probiotics in First the Trimester of Pregnancy. A Prospective Pilot Study
Brief Title: Microbiome Vaginae After Use of Oral Probiotics in Pregnancy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associate Prof. Ljubomir Petricevic MD (Other)
Responsible Party: Sponsor-Investigator, Associate Prof. Ljubomir Petricevic MD, principal investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP2021/INF1.1
Record Dates: First submitted 2021-02-23; First posted 2021-03-03 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Pregnancy; Infection Genitourinary System
Keywords: probiotics; pregnant women; microbiome
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Receiving Oral Probiotics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic group (Experimental): pilot study with one interventional group
  Interventions: Dietary Supplement: Oral probiotics

INTERVENTIONS:
Dietary Supplement: Oral probiotics — containing four Lactobacillus strains (Lactobacillus crispatus -Lbv88, Lactobacillus rhamnosus -Lbv96, Lactobacillus jensenii -Lbv116, and Lactobacillus gasseri -Lbv150)

SUMMARY:
Change of Vaginal microbiome in first trimester pregnant women after oral intake of Probiotic preparation with 4 lactobacilli strains

DETAILED DESCRIPTION:
Although the research of the vaginal microbiome is taking faster pace in recent years than it was the case before, there is still lack of information, about its composition, how and when it changes and how that can affect processes in the female body.

During pregnancy, the microbiome physiologically gets increasingly stable. Diversity of bacteria decreases, which is the sign of a healthy microbiome, and Lactobacillus species increase their already pre-existing dominance. Acidic metabolites of those bacteria maintain the low pH and low diversity in vagina.

If the dominance of lactobacilli is not as large as it should be, the risk of preterm birth increases significantly. Low relative abundance of Lactobacillus species, especially Lactobacillus crispatus (marker of the healthy microbiome) and lactobacillus metabolites as well as high vaginal microbial diversity are most significantly connected with preterm birth.

Despite such a high relevance of vaginal microbiome for a healthy pregnancy, and for women's health in general, there's an insufficient proof that the intake of oral probiotics can change it. The aim of our study is to see if the intake of patented dietary supplement, containing four Lactobacillus strains can change the relative abundance of different bacteria in the vaginal microbiome. This could lay ground for further research in this area and even create new therapeutic approaches in the future.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged between 18 and 45
* infection screening during a prenatal consultation between 10+0 (10 weeks plus 0 days) and 16+0 (16 weeks plus 0 days) gestational weeks
* Singleton pregnancy

Exclusion Criteria:

* Vaginal infections such as Bacterial vaginosis, candida vaginitis, trichomoniasis, mycoplasma, gonococcal infection
* Antibiotic therapy in the last 4 weeks
* Probiotic therapy in the last 4 weeks
* Operation on gastrointestinal tract
* Diarrhoea, obstipation
* Vaginal bleeding
* Patients with hormone disorders of any kind
* Other chronic diseases (Diabetes, Autoimmune diseases etc.)
* HIV
* Gestational diabetes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — First trimester Pregnant women
Enrollment: 44 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
CST | 14 Days
  change of vaginal microbiome after probiotic intake

SECONDARY OUTCOMES:
Lactobacilli Change | 14 Days
  change of relative abundances of each Lactobacillus species contained in the probiotic

CONTACTS AND LOCATIONS:
Overall Officials: Ljubomir Petricevic, Prof Dr, Principal Investigator — Medical University Vienna
Locations (1):
- Department of Obstetrics and Gynecology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No